CLINICAL TRIAL: NCT02943655
Title: Combined Oral Contraceptives, Progestogens, and Non-steroidal Anti-inflammatory Drugs for Heavy and/or Prolonged Menstrual Bleeding Without Organic Cause
Brief Title: Treatment of Heavy and/or Prolonged Menstrual Bleeding Without Organic Cause
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HVB
Record Dates: First submitted 2016-10-21; First posted 2016-10-25 (Estimated); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Improve Quality of Life; Heavy Menstrual Bleeding
MeSH Terms: conditions — Menorrhagia | interventions — Medroxyprogesterone Acetate; Progest; Mefenamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- combined oral contraceptives (Active Comparator): oral second generation pills one tablet daily
  Interventions: Drug: combined contraceptive pills (microcept)
- medroxyprogesterone acetate (Active Comparator): oral 5 mg daily
  Interventions: Drug: medroxyprogesterone acetate (progest)
- non-steroidal anti-inflammatory (Active Comparator): oral 500 mg mefenamic acid three times per day
  Interventions: Drug: mefenamic acid (ponstan forte)

INTERVENTIONS:
Drug: combined contraceptive pills (microcept) — oral combined contraceptive once daily
  Other Names: microcept
  Arms: combined oral contraceptives
Drug: medroxyprogesterone acetate (progest) — oral 5 mg medroxyprogesterone acetate daily
  Other Names: progest
  Arms: medroxyprogesterone acetate
Drug: mefenamic acid (ponstan forte) — oral 500 mg mefenamic acid three times per day
  Other Names: ponstan forte
  Arms: non-steroidal anti-inflammatory

SUMMARY:
Abnormal uterine bleeding encompasses abnormalities in the regularity, duration of flow, frequency, and/or blood flow volume relative to normal menstruation. Of these menstrual abnormalities, heavy menstrual bleeding (HMB), defined objectively as a blood loss of 80 ml or more per menstrual cycle , which is unrelated to pregnancy or known pelvic or systemic disease.

ELIGIBILITY:
Inclusion Criteria:

Regular menstrual cycles with BMI (19-29 kg/m2). Heavy and/or prolonged menstrual bleeding involving at least last three consecutive menstrual cycles.

Exclusion Criteria:

1. Postmenopausal bleeding (over one year since the last menstrual period).
2. Irregular menses or intermenstrual bleeding.
3. Organic causes of heavy menstrual bleeding suspected or confirmed by experienced abdominal and transvaginal ultrasound after thorough general and gynecological examination.
4. Iatrogenic (treatment-related) causes of heavy menstrual bleeding (e.g. non-progestogen-releasing intrauterine contraceptive device, oral contraceptives, other hormonal drug use or anticoagulant agent).
5. Iron deficiency anemia.
6. History of chronic diseases known to interfere with menstrual bleeding or prevent the use of any of the listed drugs e.g previous or current thromboembolic disease.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
the amount of menstrual blood loss | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided